CLINICAL TRIAL: NCT05272982
Title: Thoracic Fluid Content by Electrical Cardiometry Versus Lung Ultrasound Score as Predictors of Weaning Outcome in Mechanically Ventilated Intensive Care Patients
Brief Title: Thoracic Fluid Content by Electrical Cardiometry Versus Lung Ultrasound in Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Esraa Rabie Amer, Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Tanta University
Other Study IDs: 35237/1/22
Record Dates: First submitted 2022-02-14; First posted 2022-03-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Thoracic Fluid Content; Electrical Cardiometry; Lung Ultrasound; Mechanical Ventilation; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful weaning group: Criteria of weaning included resolution of the primary cause of intubation, adequate cough without excessive tracheobronchial secretions, PaO2 > 60 mmHg with positive end-expiratory pressure ≤ 8 cmH2O, fraction of inspired oxygen ≤ 0.4, respiratory rate < 30 per minute, appropriate pH for patients' baseline respiratory status, and stable cardiovascular status.
  Interventions: Diagnostic Test: Thoracic fluid content by electrical cardiometry group; Diagnostic Test: Ultrasound examination group
- Failed weaning group: Weaning failure will be defined as a patient need for reintubation or noninvasive ventilation within 48 h after extubation due to the presence of one or more of the following criteria: altered mental status tachypnea (respiratory rate more than 35 breaths per minute), oxygen saturation less than 90% or PaO2 less than 60 mmHg on a fraction of inspired oxygen of 40%, an apparent increase in accessory respiratory muscle activity, evident facial signs of respiratory distress and hemodynamic instability (Heart rate >140 b/min, systolic blood pressure >180 or < 90mmHg )
  Interventions: Diagnostic Test: Thoracic fluid content by electrical cardiometry group; Diagnostic Test: Ultrasound examination group

INTERVENTIONS:
Diagnostic Test: Thoracic fluid content by electrical cardiometry group — Thoracic fluid content will be measured using electrical cardiometry device (ICON ® Cardiotronics, Inc., La Jolla, CA 92307; Osyka Medical GmbH, Berlin, and Germany, model C3, Serial no: 1725303). The ICON device will be connected to four electrocardiogram electrodes which will be placed over patients' skin after cleaning with alcohol at the neck below the left ear, just above the left clavicular midpoint, and two electrodes at left mid-axillary line one at the level of the xiphoid process, and the other electrode 5 cm below this point. The thoracic fluid content will be observed for 30 s and the average of the highest and lowest values will be recorded.
Diagnostic Test: Ultrasound examination group — The 12-region technique for lung assessment will be performed using Philips ® (CX50 - Extreme edition) equipped with phased array transducer. B-line will be defined as laser like vertical hyperechoic artefact which extends between the pleural line and the bottom of the screen and moves with respiratory movements. Two types of B-lines will be evaluated.

SUMMARY:
This study aims to compare the accuracy of the total thoracic fluid content (TFC) measured by electrical cardiometry with accuracy of lung ultrasound score in prediction of weaning outcome in mechanically ventilated patients.

DETAILED DESCRIPTION:
Weaning of patients from mechanical ventilation remains one of the critical decisions in the intensive care unit. Earlier patient weaning from mechanical ventilation is recommended to avoid complications of prolonged mechanical ventilation; however, premature weaning might result in extubation failure which is, independently, associated with poor outcomes.

Screening for eligibility is the first step in the weaning process, followed by the spontaneous breathing trial (SBT). Various indices should be checked carefully before starting a spontaneous breathing trial to ensure adequate oxygenation, ventilation, and airway reflexes. However, nearly one-third of patients fail and are reintubated despite fulfillment of all the current weaning pre-requisites.

ELIGIBILITY:
Inclusion Criteria:

* 85 mechanically ventilated patients for ≥ 48 hours
* Aged 18-65 years
* Both sex
* Fulfilled the weaning readiness criteria
* Scheduled for spontaneous breathing trial (SBT) using pressure support ventilation.

Exclusion Criteria:

* Acute respiratory distress syndrome (ARDS) patients.
* Interstitial lung fibrosis.
* Patients with lung resection.
* Pulmonary embolism.
* Patients with fluid overload due to heart, renal or hepatic failure.
* Cardiac patients with ejection fraction less than 40%, cardiomyopathy, congenital or valvular heart diseases.
* Pneumothorax.
* Pleural or pericardial effusion.
* Pregnancy.
* Patients with injuries, burns, or wounds which precluded the proper application of the device electrodes or the ultrasound transducer.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 85 mechanically ventilated patients for ≥ 48 hours aged 18 years or more of both sex who fulfilled the weaning readiness criteria and scheduled for spontaneous breathing trial using pressure support ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Comparing the area under the curve (AUC) of receiver operating characteristic (ROC) for thoracic fluid content (TFC) and lung ultrasound score. | Two days after the extubation
  Comparing the area under the curve (AUC) of receiver operating characteristic (ROC) for thoracic fluid content (TFC) and lung ultrasound score (minimum score, normal lungs: 0; maximum score, both consolidated lungs: 36) in prediction of weaning outcome in mechanically ventilated patients.

SECONDARY OUTCOMES:
Prediction of weaning through rapid shallow breathing index (RSBI) | Two days after the extubation
  Rapid shallow breathing index (RSBI) [respiratory rate/tidal volume (in liters)] will be recorded before the initiation of spontaneous breathing trial (SBT) and before extubation.
The degree of lung compliance | Before initiation of spontaneous breathing trial and before extubation.
  Lung compliance will be recorded before initiation of spontaneous breathing trial and before extubation.
  It is defined as the measure of the lung's ability to stretch and expand (distensibility of elastic tissue) and is calculated using the equation (V/ΔP; where ΔV is the change in volume, and ΔP is the change in pleural pressure.
Cumulative fluid balance | within 24 hours of spontaneous breathing trial
  Cumulative fluid balance at the day of spontaneous breathing trial (equals the total fluid intake minus the fluid output) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia Governorate, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: The data will be available after the study and for 5 years after.